CLINICAL TRIAL: NCT05715034
Title: Pilot Randomized Trial of Compassionate Care: A Single-Session Web-Based Training in Self-Compassion Among Adults With Stress, Anxiety, and/or Depressive Symptoms
Brief Title: Single-Session Web-Based Training in Self-Compassion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000033574
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Stress; Anxiety; Depression
Keywords: Randomized controlled trial; Self-Compassion
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compassionate Care (Experimental): Single-session, self-guided web-based intervention (~45 minutes) hosted on Qualtrics with animated videos, audio-guided exercises, graphics, text-based material, and interactive questions. This intervention is designed to teach participants about mindfulness and self-compassion.
  Interventions: Behavioral: Compassionate Care
- Relaxing with Nature (Active Comparator): Single-session self-guided web-based intervention (~30 to 45 minutes) hosted on Qualtrics with videos (real-life images), text-based material, and questions. Each video includes a sequence of pleasant nature photos (shown about 6 seconds each) with relaxing music in the background.
  Interventions: Behavioral: Relaxing with Nature

INTERVENTIONS:
Behavioral: Compassionate Care — Single-session web-based program
  Arms: Compassionate Care
Behavioral: Relaxing with Nature — Single-session web-based program
  Arms: Relaxing with Nature

SUMMARY:
Two-arm, parallel group randomized clinical trial conducted via Mturk comparing a single-session web-based intervention called Compassionate Care versus a control intervention (nature videos with relaxing music) for adults with moderate-to-severe stress, depression and/or anxiety symptoms.

DETAILED DESCRIPTION:
Procedures include completing: (1) pre-intervention baseline assessment; (2) one of two single-session web-based intervention (approximately 30 to 45 minutes each); (3) a brief post-intervention survey; and (4) a 2-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English
* At least moderate stress, anxiety and/or depressive symptoms, as indicated by a score of:

  14 or higher on the PSS-10, and/or 10 or higher on the GAD-7, and/or 10 or higher on the PHQ-9

Exclusion Criteria:

* Fail to meet above-listed inclusion criteria
* Do not pass attention/data quality checks in initial screening or study assessments, including:
* Obvious lack of English fluency in open response questions
* Responding with random text in open response questions
* Respond with either copy/pasted responses from text earlier in the intervention to any of free response questions
* Participants with a completion time less than an average of 1.5 seconds per question for the baseline survey assessment OR who fail all three attention check questions in the baseline survey, indicating very careless, random, inattentive and/or hasty responding
* Exit the study prior to condition randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change in Stress symptoms | Baseline to 2-week follow-up
  Perceived Stress Scale (PSS-10). Total scores range from 0 to 40 with higher scores indicating greater stress symptoms
Change in Anxiety symptoms | Baseline to 2-week follow-up
  General Anxiety Disorder-7 (GAD-7). Total scores range from 0 to 21, with higher scores indicating greater anxiety symptoms.
Change in Depressive symptoms | Baseline to 2-week follow-up
  Patient Health Questionnaire-9 (PHQ-9). Total scores range from 0 to 27, with higher scores indicating greater depressive symptoms.
Change in Functional Impairment | Baseline to 2-week follow-up
  Work and Social Adjustment Scale (WSAS). Total scores range from 0 to 40, with higher scores indicating greater functional impairment.

SECONDARY OUTCOMES:
Change in Self-Compassion | Baseline to 2-week follow-up
  Self-Compassion Scale (SCS). Total scores are the average of each of the subscales, and range from 0 to 5. Higher scores indicate greater self-compassion.
Change in Mindfulness | Baseline to 2-week follow-up
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Total scores range from 0 to 40, with higher scores indicating greater mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with HIPAA and Yale Human Investigation Committee standards, any data sets that will be shared will not include any personally identifiable information. Requests for data sharing will be considered within the context of ongoing and planned research being performed within the research group at Yale in order to avoid duplication of effort and overlap in data analysis that might compromise communication of findings. Data to be shared will be de-identified and transmission electronically and securely, as we have done previously with investigators at other institutions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code